CLINICAL TRIAL: NCT06432894
Title: Performance Evaluation of Analgesia Nociception Index (ANI) in Patients Under General Anaesthesia With Remimazolam: a Prospective Observational Study
Brief Title: Performance Evaluation of ANI in Patients Under General Anesthesia With Remimazolam
Status: Recruiting | Type: Observational
Sponsor: Catholic Kwandong University (Other)
Responsible Party: Principal Investigator, Jungmin Lee, Assistant Professor, Catholic Kwandong University
Other Study IDs: Ilsan_Cha_2023-04-003-005
Record Dates: First submitted 2024-05-17; First posted 2024-05-29 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Pain Measurement
Keywords: Remimazolam; Remifentanil; Analgesia Nociception Index (ANI)
MeSH Terms: interventions — remimazolam

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation: Patients
  * aged 20-80 years under general anaesthesia with remimazolam
  * scheduled to undergo robotic surgery
  * in American Society of Anesthesiologists physical class 1, 2 or 3
  Interventions: Combination Product: Analgesia Nociception Index, remimazolam

INTERVENTIONS:
Combination Product: Analgesia Nociception Index, remimazolam — The purpose of this study is to determine the validity of ANI in patients undergoing surgery with remifentanil and remimazolam.
  During this study, remimazolam infusion rate is determined by the pharmacopoeia.
  Remifentanil infusion rate is determined based on the patient's vital signs, systemic status and pain levels. And remifentanil is administrated via targeted infusion control using the Minto model.
  ANI scores, vital signs, remifentanil infusion rate are collected at predetermined time points according to the protocol from the start to the end of the surgery.

SUMMARY:
The purpose of this study is to determine whether Analgesia Nociception Index (ANI) can effectively reduce the dose of opioid in patients who underwent general anesthesia using remimazolam.

ELIGIBILITY:
Inclusion Criteria:

Patients

* aged 20-79 years under general anaesthesia with remimazolam
* scheduled to undergo robotic surgery
* in American Society of Anesthesiologists physical class 1, 2 or 3
* voluntarily agree in writing to participate in this clinical study

Exclusion Criteria:

* Conditions affecting the autonomic nervous system
* other conditions or disease that may cause acute or chronic pain
* the NRS before induction of anesthesia is 1 or over
* When taking medications that may affect the autonomic nervous system
* In other cases where the investigator deems the subject unsuitable for this trial

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who visit the hospital and undergo surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2025-06-11 (Estimated); Study Completion 2025-06-11 (Estimated)

PRIMARY OUTCOMES:
ANI values | During Surgery (at the points of intubation, skin incision, CO2 insufflation, TOF stimulation, and hemodynamic change)
  A value indicating the degree of pain calculated by ANI's algorithm

SECONDARY OUTCOMES:
Heart Rate (HR) change | Every 2 seconds for 2.5 minutes before and Every 2 seconds for 2.5 minutes after pain stimulation
  Because the ANI value is calculated using the change in HR, it is measured to correlate the change in ANI value with the change in HR due to pain.
Patient state index (PSI) change | Every 2 seconds for 2.5 minutes before and Every 2 seconds for 2.5 minutes after pain stimulation
  The PSI is an indicator of a patient's depth of sedation and is calculated based on EEG, which can change in response to painful stimuli. The PSI score is expressed as a number between 0 and 100, and it is usually recommended to maintain under 60 during surgery. An increase in the PSI score can indicates the degree of pain stimulus and can be used as an indicator to assess the validity of the ANI value.
Blood Pressure change | Every 2 seconds for 2.5 minutes before and Every 2 seconds for 2.5 minutes after pain stimulation
  When a patient feels pain, it stimulates the autonomic nervous system to change blood pressure. This change is measured to determine how much pain the patient is feeling
Remimazolam infusion rate | During Surgery (at the points of intubation, skin incision, CO2 insufflation, TOF stimulation, and hemodynamic change)
  Remimazolam is a sedative. The infusion rate of remimazolam correlates with sedation level. And it is measured to determine if sedation level correlates with ANI values when pain stimuli are given.
Effect site concentration of remifentanil | During Surgery (at the points of intubation, skin incision, CO2 insufflation, TOF stimulation, and hemodynamic change)
  Remifentanil is an opioid and can affect pain levels when given a pain stimulus.

OTHER OUTCOMES:
Hemodynamic change | within 5 minutes of pain stimulus
  When there are changes of heart rate or blood pressure more than 20% from baseline within 5 minutes of pain stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Young Joo, Study Chair — Ilsan Cha hospital
Locations (1):
- Catholic-Kwandong University, School of Medicine, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code